CLINICAL TRIAL: NCT00641927
Title: Acute Antidepressant Therapy in Bipolar II Major Depression
Brief Title: Antidepressant Therapy for Bipolar II Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanley Medical Research Institute (Other)
Responsible Party: Jay D. Amsterdam, MD, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-005
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Bipolar Type II Disorder
Keywords: bipolar disorder; bipolar type II disorder; antidepressant; mood stabilizer; venlafaxine; lithium carbonate
MeSH Terms: conditions — Bipolar Disorder | interventions — Venlafaxine Hydrochloride; Lithium Carbonate; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Antidepressant
  Interventions: Drug: Venlafaxine
- 2 (Active Comparator): Drug
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Venlafaxine — 37.5 mg - 375 mg daily, 12 Weeks
  Other Names: Effexor-XR
  Arms: 1
Drug: Lithium Carbonate — 300 mg - 2100 mg daily, 12 weeks
  Other Names: Lithium
  Arms: 2

SUMMARY:
This study examines the relative safety and benefit of antidepressant therapy (versus recommended mood stabilizer therapy)of bipolar type II major depressive episode. We hypothesize that antidepressant therapy will be superior to mood stabilizer therapy with little or no difference in treatment emergent manic symptoms.

DETAILED DESCRIPTION:
Bipolar type II (BP II) major depressive episode (MDE), affects 2.5% of the US adult population and results in an estimated healthcare cost of $40 billion annually. BP II disorder is a distinct clinical entity that differs from BP I disorder, and is characterized by a preponderance of MDEs that result in particularly high morbidity and mortality rates. The treatment of BP II MDE remains a challenge for clinicians. Concerns over antidepressant drug (AD) induced manic switch episodes have led current practice guidelines to recommend treating BP II MDE with mood stabilizer (MS) monotherapy and to avoid AD monotherapy. To date, there are no controlled clinical trials to test the validity of these empirical guidelines. Results from our preliminary BP II MDE studies have shown that fluoxetine monotherapy may be safe and effective initial treatment of BP II MDE with a low manic switch rate. Based upon these observations, we now ask (Specific aim #1): "What is the relative safety and efficacy of initial AD monotherapy vs. MS monotherapy of BP II MDE?" and "What is the relative manic switch rate of initial AD vs. MS monotherapy of BP II MDE?" To answer these questions, patients with BP II MDE will be treated in a 12-week, randomized, parallel group comparison of venlafaxine monotherapy vs. lithium monotherapy. We hypothesize that AD monotherapy will have superior efficacy vs. MS monotherapy, and that there will be a similar manic switch rate among both treatment conditions. If our hypotheses are correct, we believe that these results may have an important public health impact on the current practice guidelines for treating BP II MDE.

ELIGIBILITY:
Inclusion Criteria:

* men and women (all races and ethnicity) greater than or equal to18 years of age,
* DSM IV diagnosis of BP II disorder,
* Current DSM IV MDE,
* HAM-D17 score greater than or equal to 16,
* Drug free from prior psychotropic medication greater than or equal to 7 days (2 weeks for MAOIs)

Exclusion Criteria:

* History of mania,
* Other primary DSM IV Axis I diagnosis,
* Alcohol or drug dependence within 3 months,
* History of nonresponse to Effexor-XR or lithium in the present MDE,
* History of allergic reaction to Effexor-XR or lithium,
* Medical contraindications to treatment with Effexor-XR or lithium,
* Unstable medical condition,
* Pregnant or breast-feeding women,
* Women of child-bearing potential not using a medically approved form of contraception,
* Actively suicidal or requiring hospitalization,
* Requiring concurrent antidepressant, neuroleptic or mood stabilizer therapy,
* Prior investigational study within 4 weeks of starting active therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Reduction in Hamilton Depression Rating Scale score. | 12 Weeks

SECONDARY OUTCOMES:
Change in Young Mania Rating Scale score. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay D Amsterdam, MD, Principal Investigator — Depression Research Unit, School of Psychiatry, University of Pennsylvania
Locations (1):
- Depression Research Unit, Department of Psychiatry, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Shults J, Sun W, Tu X, Kim H, Amsterdam J, Hilbe JM, Ten-Have T. A comparison of several approaches for choosing between working correlation structures in generalized estimating equation analysis of longitudinal binary data. Stat Med. 2009 Aug 15;28(18):2338-55. doi: 10.1002/sim.3622. PMID 19472307